CLINICAL TRIAL: NCT04471948
Title: The Safety and Efficacy of 1064-nm Picosecond Laser 1064 With Microlens Array for Pore Tightening; a Pilot Study
Brief Title: The Safety and Efficacy of 1064-nm Picosecond Laser With Microlens Array for Pore Tightening; a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si379/2019
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Enlarged Pores
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fractional picosecond laser 1,064 nm laser (Experimental): 1 arm The subjects with enlarged pores were treated with fractional picosecond laser 1,064 nm laser
  Interventions: Device: Fractional picosecond 1064 nm laser

INTERVENTIONS:
Device: Fractional picosecond 1064 nm laser — The parameter of laser was 8 mm spot size, 0.8 mJ/CM2, 750 ps, 5 Hz, 2 passes The treatment was done in every 4 weeks for 3 sessions.

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of 1064-nm Picosecond laser 1064 With Microlens Array for Pore tightening.

DETAILED DESCRIPTION:
The Safety and Efficacy of Picosecond laser 1064 Nanometers With Microlens Array for Pore tightening; a Pilot Study Primary outcome : pore size Secondary outcome : side effect, patient satisfaction, global evaluation the patient recieved laser treament once a month for 3 months and then follow up after last treatment at 1, 3 ,6 month

Enlarged facial pores is one of the skin signs in photoaging. There are 3 major clinical causes of enlarged facial pores: highs sebum excretion, decreased elasticity around pores and increased hair follicle volume. Possible causative factors of enlarged facial pores include many exogenous and endogenous factors include genetic predisposition, seborrhea and chronic ultraviolet light exposure. Picosecond laser are new device which has been used in skin rejuvenation. The main mechanism of action is laser induced optical breakdown (LIOB).

ELIGIBILITY:
Inclusion Criteria:

* Both male and female age 25-40 years
* No underlying disease

Exclusion Criteria:

* History of retinoid or other keratolytic drugs used within 6 months before enrolled
* History of keloid
* photosensitivity
* Immunocompromised host

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-03-07 (Estimated); Study Completion 2021-03-07 (Estimated)

PRIMARY OUTCOMES:
Change in pore size by Antera 3D image | change from baseline in pore size at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: woraphong Manuskiatti, M.D., Principal Investigator — Mahidol University
Locations (1):
- Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Thailand